CLINICAL TRIAL: NCT05439135
Title: An Open-label, Multicenter, Randomized Clinical Trial for Malnutrition After Nonphysiological Reconstruction of the Upper Gastrointestinal Tract: Washed Microbiota Transplantation Via Mid-gut Tube Versus Colonic Transendoscopic Enteral Tube
Brief Title: Washed Microbiota Transplantation for Malnutrition After Nonphysiological Reconstruction of the Upper Gastrointestinal Tract
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: The First Affiliated Hospital of Guangdong Pharmaceutical University (Other); Nanjing Medical University (Other); Wuxi No. 2 People's Hospital (Other); Jiangxi University of Chinese Medicine Affiliated Hospital (Unknown); Hubei Hospital of Traditional Chinese Medicine (Other); The Affiliated Hospital Of Southwest Medical University (Other); Tang-Du Hospital (Other); Huzhou Central Hospital (Other); West China Forth University Hospitalï¼ŒSichuan University (Unknown); The Affiliated People's hospital of Ningbo Univercity (Other); Guangzhou First People Hospital of Guangzhou Medical University (Unknown); The First Affiliated Hospital of Anhui University of Chinese Medicine (Other); Beijing Rectum Hospital (Unknown); Dazhou Central Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); The 901th Hospital of Joint Logistics Support Force of Chinese People's Liberation Army (Unknown); YI'AN PEOPLE'S HOSPITAL (Unknown); Hunan Aerospace Hospital (Unknown); Jiamusi City Hospital of Traditional Chinese Medicine (Unknown); The First People's Hospital of Kunshan (Other); LanZhou University (Other); Jingxing xian yiyuan (Unknown); TAIHE country people's hospital (Unknown); Tailai County People's Hospital (Unknown); Armed Police Characteristic Medical Center (Unknown); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Associate professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DELIV2022N002
Record Dates: First submitted 2022-06-19; First posted 2022-06-30 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2024-10

CONDITIONS: Malnutrition; Gastroenterostomy
Keywords: washed microbiota transplantation; fecal microbiota transplant; malnutrition; enteral nutrition; cachexia; upper gastrointestinal rerouting surgery; delivery; nonphysiological reconstruction of the upper gastrointestinal tract
MeSH Terms: conditions — Malnutrition; Cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- midgut (Experimental): A soft TET tube is inserted into the colon via the paraffin-lubricated gastroscope channel. If patients cannot tolerate endoscopy or anesthesia, or it is difficult to confirm the bypass intestine under endoscopy, a nasojejunal tube will be inserted under digital fluoroscopy.
  Interventions: Other: washed microbiota transplantation
- colonic (Experimental): A soft TET tube is inserted into the colon via the paraffin-lubricated colonoscope channel.
  Interventions: Other: washed microbiota transplantation

INTERVENTIONS:
Other: washed microbiota transplantation — Each patient will receive washed microbiota transplantation each day for three consecutive days. After WMT, participants will receive free diet plus home enteral nutrition (solution at a 750ml daily dosage that provides 750 kcal energy) at home for 8 weeks.
  Other Names: home enteral nutrition

SUMMARY:
This is a prospective, randomized, multicenter study to evaluate WMT in improving nutritional status in malnourished patients who underwent nonphysiological reconstruction of the upper gastrointestinal tract. In this multicenter trial, sixty-two patients will be enrolled in forteen Chinese sites. Participants will be randomized at a ratio of 1:1 to receive three WMTs through either mid-gut tube or colonic TET. After WMT, each participant will receive free diet plus home enteral nutrition. Home enteral nutrition should last for 2 months at home, with blood, urine and stool samples taken and stored at baseline and 2 months after WMT.

DETAILED DESCRIPTION:
Background: Malnutrition is a common complication of nonphysiological reconstruction of the upper gastrointestinal tract. The potential of washed microbiota transplantation (WMT) in improving nutritional status have been reported. The surgery procedure alters the anatomy and physiology of the digestive tract, which might impact the efficacy and safety of WMT when choosing different delivery way. This study aims to explore the optimal delivery of WMT in malnourished patients after rerouting of the upper gastrointestinal tract.

Methods and design: This multicenter, open-label, and randomized controlled trial will be conducted at forteen hospitals in China. Enteral nutrition (EN) will be administrated at enrollment. Participants will be then randomized at a ratio of 1:1 to receive three WMTs through either mid-gut tube or colonic transendoscopic enteral tubing (TET). Then the patients will receive free diet coupled with home enteral nutrition (HEN) for 8 weeks in both groups, with blood, urine and stool samples taken and stored at baseline and 2 months after WMT. The observation duration is 8 weeks. The primary endpoint is nutritional status of the patients. The nutritional status data obtained at baseline and 8 weeks after discharge includes body mass index (BMI) and skeletal muscle index (SMI). The secondary endpoints are nutritional assessment, nutrition-based laboratory indices, 60-day readmission rate, quality of life, gastrointestinal symptom scale, the safety of WMT and further analysis of the biological specimens.

Conclusion: It is estimated that WMT would help improve nutrition status. Moreover, this trial has the potential to identify the optimal delivery of WMT for patients undergoing nonphysiological reconstruction of the upper gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone nonphysiological reconstruction of the gastrointestinal tract (such as Billroth-II, Roux-en-Y, Child, Whipple reconstruction)
* Aged over 18 years old;
* Malnutrition is assessed by Nutritional Risk Screening 2002 score≥3 and Patient Generated Subjective Global Assessment (PG-SGA) score≥4;
* Written informed consent;

Exclusion Criteria:

* Expected survival time < 3 months;
* Still on anti-tumor therapy or it is expected during the visit;
* Complicated with ascites or edema caused by malnutrition;
* Known organic gastrointestinal disease (e.g., gastrointestinal infection, inflammatory bowel disease, or radiation enteritis);
* Undergone other gastrointestinal surgery (e.g., enterectomy, enterostomy, or gastrostomy) except appendectomy or anal fistula surgery;
* Complicated with contraindications of enteral nutrition such as ileus, active gastrointestinal bleeding, and shock;
* Cannot tolerate gastroscopy or colonoscopy;
* Severe comorbidities (e.g., diabetes, cardiopulmonary failure, severe liver or or kidney diseases);
* Complicated with other wasting diseases (e.g., active tuberculosis, hyperthyroidism, diabetes, HIV, active hepatitis, hip fracture, craniocerebral injury, etc.);
* A history of anti-infective treatment within 30 days before enrollment; or need anti-infective treatment at the time of enrollment; or unwilling to stop taking drugs that affect gut microbes, such as probiotics;
* Can not tolerate oral enteral nutrition;
* Women who are pregnant or breastfeeding;
* Participating in another clinical trial;
* Deemed unsuitable for inclusion by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes of weight and height | baseline, 8 weeks post transplantation
  Weight and height will be combined to report BMI in kg/m^2.
Changes of the third lumbar vertebrae skeletal muscle mass and height | baseline, 8 weeks post transplantation
  The third lumbar vertebrae skeletal muscle mass represents the sum of the cross-sectional areas of the skeletal muscles at the L3 level, including the psoas major, the erector spinae, the quadratus lumborum, the musculus transversus abdominis, the obliquus externus abdominis and the obliquus internus abdominis. Skeletal muscle mass and height will be combined to report the third lumbar vertebrae skeletal muscle mass index(L3 SMI) in cm^2/m^2.
Changes of weight | baseline, 8 weeks post transplantation

SECONDARY OUTCOMES:
Changes of Patient-Generated Subjective Global Assessment (PG-SGA) | baseline, 8 weeks post transplantation
  Patient-Generated Subjective Global Assessment (PG-SGA) includes patient-generated historical components (Weight History, Food Intake, Symptoms and Activities and Function) and the professional part (Diagnosis, Age, Metabolic stress, and Physical Exam).
Changes of the Gastrointestinal Symptom Rating Scale(GSRS) | baseline, 4 weeks, 8 weeks post transplantation
  GSRS is a 13-item test to make a comprehensive assessment of common gastrointestinal symptom and each item receives a value from 0 to 3, with higher value indicating worse gastrointestinal condition.
60-day readmission rate | From enrollment to the end of treatment at 8 weeks
  The 60-day readmission is recorded and defined as nonelective readmission within 60 days after the treatment.
The incidence of treatment-related adverse events (AE) assessed by CTCAE, Version 5.0 | From enrollment to the end of treatment at 8 weeks
  The severity of AE was graded as mild (grade 1), moderate (grade 2), severe/disabling (grade 3), life threatening (grade 4), and death (grade 5). All AE were divided in definitely, probably and possibly related to treatment. The treatment-related AE we focused on included microbiota-related AEs (e.g., infection, diarrhea, abdominal pain, etc.) and route of delivery related AEs (e.g., nausea, vomiting, etc.).
Changes of the 5-level EuroQoL Group's 5-dimension (EQ-5D-5L) | baseline, 4 weeks, 8 weeks post transplantation
  EQ-5D-5L is a 5-dimension questionnaire measuring health state and each dimension represents the level from 1 to 5, with higher level indicating worse health state.
Changes of the Pittsburgh Sleep Quality Index (PSQI) | baseline, 4 weeks, 8 weeks post transplantation
  PSQI is a self-rated questionnaire which assesses sleep quality over a 1-month time interval. Nineteen items generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for seven components yields one global score, with higher score indicating worse sleep quality.
Changes of the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) | baseline, 4 weeks, 8 weeks post transplantation
  FACIT-Fatigue is a 13-item test measuring fatigue and each item receives a value from 0 to 4, with higher value indicating worse fatigue state.
The difference of the gut microbiota composition before and after washed microbiota transplantation | baseline, 8 weeks post transplantation
  The composition of the gut microbiota is evaluated by sequencing faecal metagenome. We evaluate the differences in the structure of the flora and its metabolism.
Change of insulin-like growth factor I(IGF-I) | baseline, 8 weeks post transplantation
  Blood is tested for Insulin-like growth factor I.
Changes of hemoglobin | baseline, 8 weeks post transplantation
  Blood is tested for hemoglobin
Changes of albumin | baseline, 8 weeks post transplantation
  Blood is tested for albumin
Changes of prealbumin | baseline, 8 weeks post transplantation
  Blood is tested for prealbumin
Changes of cholesterol | baseline, 8 weeks post transplantation
  Blood is tested for cholesterol
Changes of transferrin | baseline, 8 weeks post transplantation
  Blood is tested for transferrin
Changes of C-reactive protein | baseline, 8 weeks post transplantation
  Blood is tested for C-reactive protein
Changes of full spectrum of bile acidsare | baseline, 8 weeks post transplantation
  Blood is tested for full spectrum of bile acidsare, including Cholic acid, deoxycholic acid, chenodeoxycholic acid, urs/hyodeoxycholic acid, lithocholic acid, glycocholic acid, glycolithocholic acid, glycodeoxycholic acid, glycochenodeoxycholic acid, glycouran Deoxycholic acid, taurocholic acid, taurolithocholic acid, taurodeoxycholic acid, taurochenodeoxycholic acid, tauroursodeoxycholic acid.
Changes of glucose breath testing | baseline, 8 weeks post transplantation
  A baseline breath sample was obtained, patients drank 50g glucose dissolved in 8 ounces of water, and breath samples were obtained at 15-minute intervals for 2 hours. Samples were analyzed to calculate breath H2 and/or breath CH4.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Csendes A, Burgos AM, Smok G, Burdiles P, Braghetto I, Diaz JC. Latest results (12-21 years) of a prospective randomized study comparing Billroth II and Roux-en-Y anastomosis after a partial gastrectomy plus vagotomy in patients with duodenal ulcers. Ann Surg. 2009 Feb;249(2):189-94. doi: 10.1097/SLA.0b013e3181921aa1. PMID 19212169
- [Background] Nishizaki D, Ganeko R, Hoshino N, Hida K, Obama K, Furukawa TA, Sakai Y, Watanabe N. Roux-en-Y versus Billroth-I reconstruction after distal gastrectomy for gastric cancer. Cochrane Database Syst Rev. 2021 Sep 15;9(9):CD012998. doi: 10.1002/14651858.CD012998.pub2. PMID 34523717
- [Background] Zhang F, Luo W, Shi Y, Fan Z, Ji G. Should we standardize the 1,700-year-old fecal microbiota transplantation? Am J Gastroenterol. 2012 Nov;107(11):1755; author reply p.1755-6. doi: 10.1038/ajg.2012.251. No abstract available. PMID 23160295
- [Background] Xiang L, Yu Y, Ding X, Zhang H, Wen Q, Cui B, Zhang F. Exclusive Enteral Nutrition Plus Immediate vs. Delayed Washed Microbiota Transplantation in Crohn's Disease With Malnutrition: A Randomized Pilot Study. Front Med (Lausanne). 2021 Oct 22;8:666062. doi: 10.3389/fmed.2021.666062. eCollection 2021. PMID 34746161
- [Background] Levine A, Wine E, Assa A, Sigall Boneh R, Shaoul R, Kori M, Cohen S, Peleg S, Shamaly H, On A, Millman P, Abramas L, Ziv-Baran T, Grant S, Abitbol G, Dunn KA, Bielawski JP, Van Limbergen J. Crohn's Disease Exclusion Diet Plus Partial Enteral Nutrition Induces Sustained Remission in a Randomized Controlled Trial. Gastroenterology. 2019 Aug;157(2):440-450.e8. doi: 10.1053/j.gastro.2019.04.021. Epub 2019 Jun 4. PMID 31170412
- [Background] Peng Z, Xiang J, He Z, Zhang T, Xu L, Cui B, Li P, Huang G, Ji G, Nie Y, Wu K, Fan D, Zhang F. Colonic transendoscopic enteral tubing: A novel way of transplanting fecal microbiota. Endosc Int Open. 2016 Jun;4(6):E610-3. doi: 10.1055/s-0042-105205. Epub 2016 Apr 28. PMID 27556065